CLINICAL TRIAL: NCT03676257
Title: Survival Endpoints for Treatment Evaluation in Subjects Treated for Metastatic Breast Cancer: Contribution of Real-life Databases
Brief Title: Survival Endpoints in Women Treated for Metastatic Breast Cancer: Contribution of Real-life Databases
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Collaborators: UNICANCER (Other); Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Other Study IDs: IB-2017DATECAN-ESME
Record Dates: First submitted 2018-09-17; First posted 2018-09-18 (Actual); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic breast cancer; Real world data; Surrogate
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Women with a diagnosis of HR+ /HER2- metastatic breast cancer (mBC): Women with a diagnosis of HR+ /HER2- metastatic breast cancer (mBC)
  Interventions: Drug: Chemotherapy (exclusive); Drug: Endocrine therapy (exclusive); Drug: Combination of endocrine therapy and chemotherapy; Drug: Chemotherapy and targeted treatment; Drug: Combination of endocrine therapy and targeted treatment; Drug: Combination of chemotherapy, endocrine therapy and targeted treatment
- Women with a diagnosis of HR- /HER2- metastatic breast cancer (mBC): Women with a diagnosis of HR- /HER2- metastatic breast cancer (mBC)
  Interventions: Drug: Chemotherapy (exclusive); Drug: Chemotherapy and targeted treatment
- Women with a diagnosis of HR+ /HER2+ metastatic breast cancer (mBC): Women with a diagnosis of HR+ /HER2+ metastatic breast cancer (mBC)
  Interventions: Drug: Chemotherapy (exclusive); Drug: Endocrine therapy (exclusive); Drug: Combination of endocrine therapy and chemotherapy; Drug: Chemotherapy and targeted treatment; Drug: Combination of endocrine therapy and targeted treatment; Drug: Combination of chemotherapy, endocrine therapy and targeted treatment
- Women with a diagnosis of HR- /HER2+ metastatic breast cancer (mBC): Women with a diagnosis of HR- /HER2+ metastatic breast cancer (mBC)
  Interventions: Drug: Chemotherapy (exclusive); Drug: Chemotherapy and targeted treatment

INTERVENTIONS:
Drug: Chemotherapy (exclusive) — Administration of any chemotherapeutic agent(s)
Drug: Endocrine therapy (exclusive) — Administration of any type of endocrine therapy
  Groups: Women with a diagnosis of HR+ /HER2+ metastatic breast cancer (mBC); Women with a diagnosis of HR+ /HER2- metastatic breast cancer (mBC)
Drug: Combination of endocrine therapy and chemotherapy — Any combination of endocrine therapy and chemotherapy
  Groups: Women with a diagnosis of HR+ /HER2+ metastatic breast cancer (mBC); Women with a diagnosis of HR+ /HER2- metastatic breast cancer (mBC)
Drug: Chemotherapy and targeted treatment — Any combination of chemotherapy and targeted treatment(s)
Drug: Combination of endocrine therapy and targeted treatment — Any combination of endocrine therapy and targeted treatment
  Groups: Women with a diagnosis of HR+ /HER2+ metastatic breast cancer (mBC); Women with a diagnosis of HR+ /HER2- metastatic breast cancer (mBC)
Drug: Combination of chemotherapy, endocrine therapy and targeted treatment — Any combination of chemotherapy, endocrine therapy and targeted treatment(s)
  Groups: Women with a diagnosis of HR+ /HER2+ metastatic breast cancer (mBC); Women with a diagnosis of HR+ /HER2- metastatic breast cancer (mBC)

SUMMARY:
Overall survival (OS) is considered the most reliable cancer endpoint and used by the Health Rregulatory authorities (HRA). OS presents multiple advantages in cancer randomized controlled trials (RCT): it is universally accepted as a measure of clinical benefit for the patient; it is objectively defined, both in terms of events and date of incidence; it is easily and precisely measured and thus reproducible; it can be exhaustively collected. As such, OS has been validated by HRAs. On the other hand, OS presents some limitations. Observing a benefit on OS may require a large number of patients and/or considerable time for patient follow-up. Costs for trials may be increased, and there might be delays in the introduction of possible beneficial treatments for patients. The development of alternative endpoints that could capture treatment benefit appropriately and be measurable earlier, is central for the evolution of clinical research in oncology.

Real world data (RWD) are defined as other sources than clinical trials such as: electronic medical records, registries, insurance claims, pharmacy records, death certificates and other patient-generated data.

This research is aimed at (i) describing the existing endpoints of survival in real-life setting, (ii) comparing the correlation at individual level with data to clinical trials for related to anti-HER2 targeted therapies and endocrine therapies in MBC. We will investigate the individual correlation between candidate surrogate endpoints and overall survival in a population-based record-computerized database centralizing data on about 20,000 patients from 2008 to 2017 in France.

This work should lead to the estimation of various time-to event endpoints (e.g. OS, PFS, etc), in the real-life setting, for mBC patients. In addition, we will estimate their individual correlation with OS, which should help us highlight potential surrogate endpoints in this setting. We will focuss on three distinct population, accounting for a large population of mBS patients: : patients treated with anti-HER2 targeted agents, patients treated with endocrine therapies and elderly population.

ELIGIBILITY:
ELIGIBILITY

* female patients older than 18 years
* diagnosis of metastatic breast cancer (de novo disease or first metastatic recurrence) between January 1, 2008, and December 31, 2017
* received a fist-line systemic treatment such as chemotherapy, endocrine therapy or targeted therapy, whatever the sequence (monotherapy or combination of therapies using distinct mechanisms of actions, i.e., polytherapy).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data source : We extracted data from the ESME mBC database (NCT03275311) which gathers deidentified data from consecutive patients managed in 18 French Comprehensive Cancer Centers. Adult women diagnosed with mBC between 2008 and 2017 were included. The Epidemio-Strategy and Medical Economic (ESME) Research Program is a French academic initiative supporting the centralization of structured and non- structured data documented in the electronic health records (EHR) (clinical notes, pathology reports and radiology reports) of patients treated for malignant conditions in a unique secured web-based data platform available for researchers. The ESME mBC data platform is an EHR-derived database that gathers exhaustive data on consecutive patients who initiated a L1 treatment for mBC between 01 January 2008 and 31 December 2017 in one of 18 French Comprehensive Cancer Centers.
Sampling Method: Non-Probability Sample
Enrollment: 20033 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Insitut Bergonié, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No
Availability of data and materials : The data that support the findings of this study are available from UNICANCER but restrictions apply to the availability of these data, which were used under license for the current study, and so are not publicly available. Data are however available from the authors upon reasonable request and with permission of UNICANCER.

REFERENCES:
- [Result] Courtinard C, Gourgou S, Jacot W, Carton M, Guerin O, Vacher L, Bertaut A, Le Deley MC, Perol D, Marino P, Levy C, Uwer L, Perrocheau G, Schiappa R, Bachelot F, Parent D, Breton M, Petit T, Filleron T, Loeb A, Mathoulin-Pelissier S, Robain M, Delaloge S, Bellera C. Association between progression-free survival and overall survival in women receiving first-line treatment for metastatic breast cancer: evidence from the ESME real-world database. BMC Med. 2023 Mar 8;21(1):87. doi: 10.1186/s12916-023-02754-5. PMID 36882736
- See also: Related Info — https://www.unicancer.fr/en/programs/esme/

RESULTS

PARTICIPANT FLOW:
Groups:
- Women With a Diagnosis of HR+ /HER2- Metastatic Breast Cancer (mBC): Women with a diagnosis of HR+ /HER2- metastatic breast cancer (mBC) and satisfying eligibility criteria
- Women With a Diagnosis of HR- /HER2- Metastatic Breast Cancer (mBC): Women with a diagnosis of HR- /HER2- metastatic breast cancer (mBC) and satisfying eligibility criteria
- Women With a Diagnosis of HR+ /HER2+ Metastatic Breast Cancer (mBC): Women with a diagnosis of HR+ /HER2+ metastatic breast cancer (mBC) and satisfying eligibility criteria
- Women With a Diagnosis of HR- /HER2+ Metastatic Breast Cancer (mBC): Women with a diagnosis of HR- /HER2+ metastatic breast cancer (mBC) and satisfying eligibility criteria
Period: Overall Study
Arm/Group | Women With a Diagnosis of HR+ /HER2- Metastatic Breast Cancer (mBC) | Women With a Diagnosis of HR- /HER2- Metastatic Breast Cancer (mBC) | Women With a Diagnosis of HR+ /HER2+ Metastatic Breast Cancer (mBC) | Women With a Diagnosis of HR- /HER2+ Metastatic Breast Cancer (mBC)
Started | 13283 | 2845 | 2502 | 1403
Completed | 13283 | 2845 | 2502 | 1403
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Women With a Diagnosis of HR+ /HER2- Metastatic Breast Cancer (mBC) | Women With a Diagnosis of HR- /HER2- Metastatic Breast Cancer (mBC) | Women With a Diagnosis of HR+ /HER2+ Metastatic Breast Cancer (mBC) | Women With a Diagnosis of HR- /HER2+ Metastatic Breast Cancer (mBC) | Total
Number analyzed (Participants) | 13283 | 2845 | 2502 | 1403 | 20033
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Age at diagnosis
  years | 62 [51 to 71] | 56 [45 to 66] | 57 [47 to 67] | 56 [46 to 64] | 60 [50 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13283 | 2845 | 2502 | 1403 | 20033
  Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  France | 13283 | 2845 | 2502 | 1403 | 20033
Grade [Count of Participants; unit: Participants] — Histological grade at diagnosis. Histological grade was derived using the first informative results on the primary tumor whatever breast surgical procedures (biopsy, tumorectomy, lumpectomy, and mastectomy). Ranges from 0 (poor prognosis) to 3 (better prognosis)
  Participants
    Grade 1 | 1532 | 46 | 132 | 16 | 1726
    Grade 2 | 6883 | 758 | 1125 | 459 | 9225
    Grade 3 | 2775 | 1662 | 866 | 724 | 6027
    Grade not documented | 2093 | 379 | 379 | 204 | 3055

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) for Commonly Prescribed First-line Treatment Strategies
Description: OS was defined as the time from diagnosis of mBC to the date of death from any cause.
Time Frame: 10 years
Population: OS is reported for major combinations of treatments. For the combination of treatments "OTHER", OS is not reported given the populations are highly heterogeneous, and therefore reporting OS is not clinically relevant.
  When the number of participants in a row is "0", this means that the combinbation of treatments (defined by the row) was provided to 0 woman of the population (defined by the column).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Women With a Diagnosis of HR+ /HER2- Metastatic Breast Cancer (mBC) | Women With a Diagnosis of HR- /HER2- Metastatic Breast Cancer (mBC) | Women With a Diagnosis of HR+ /HER2+ Metastatic Breast Cancer (mBC) | Women With a Diagnosis of HR- /HER2+ Metastatic Breast Cancer (mBC)
Number analyzed (Participants) | 13268 | 2725 | 2306 | 1239
months
  Chemotherapy (exclusive): number analyzed (Participants) | 1631 | 1804 | 84 | 75
  Chemotherapy (exclusive) | 23.7 [22.2 to 25.9] | 13.5 [12.6 to 14.3] | 30.9 [23.3 to 38.7] | 17.4 [11.0 to 20.6]
  Endocrine therapy (exclusive): number analyzed (Participants) | 5545 | 0 | 342 | 0
  Endocrine therapy (exclusive) | 48.8 [47.3 to 50.2] |  | 40.3 [36.9 to 49.4] |
  Combination of endocrine therapy and chemotherapy: number analyzed (Participants) | 3383 | 0 | 85 | 0
  Combination of endocrine therapy and chemotherapy | 48.5 [46.1 to 50.3] |  | 29.5 [24.8 to 46.3] |
  Chemotherapy and targeted treatment: number analyzed (Participants) | 699 | 921 | 674 | 1164
  Chemotherapy and targeted treatment | 27.8 [25.0 to 29.9] | 15.8 [14.9 to 17.7] | 47.6 [41.3 to 55.0] | 43.8 [40.2 to 49.1]
  Combination of endocrine therapy and targeted treatment: number analyzed (Participants) | 492 | 0 | 85 | 0
  Combination of endocrine therapy and targeted treatment | 58.8 [49.5 to 69.3] |  | 56.3 [46.2 to 79.4] |
  Combination of chemotherapy, endocrine therapy and targeted treatment: number analyzed (Participants) | 1518 | 0 | 1036 | 0
  Combination of chemotherapy, endocrine therapy and targeted treatment | 42.6 [40.8 to 46] |  | 86.1 [74.5 to 97.7] |

2. Secondary Outcome: Real-world Progression-free Survival (rwPFS) for Commonly Prescribed First-line Treatment Strategies
Description: rwPFS was defined as the delay between time from initial diagnosis of mBC to the date of disease progression (regional recurrence, progression, appearance/occurrence of metastases and distant recurrence) or death (any cause), whichever came first.
  Disease progression was assessed by the treating physician based on observed clinical events, as per routine practice (regional recurrence, progression, appearance/occurrence of metastases and distant recurrence). These events were recorded in the patient medical record. As this study relates to real-world data, no specific procedure was imposed to assess these events.
Time Frame: 10 years
Population: rwPFS is reported for major combinations of treatments. For the combination of treatments "OTHER", rwPFS is not reported given the populations are highly heterogeneous, and therefore reporting rwPFS is not clinically relevant.
  When the number of participants in a row is "0", this means that the combinbation of treatments (defined by the row) was provided to 0 woman of the population (defined by the column).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Women With a Diagnosis of HR+ /HER2- Metastatic Breast Cancer (mBC) | Women With a Diagnosis of HR- /HER2- Metastatic Breast Cancer (mBC) | Women With a Diagnosis of HR+ /HER2+ Metastatic Breast Cancer (mBC) | Women With a Diagnosis of HR- /HER2+ Metastatic Breast Cancer (mBC)
Number analyzed (Participants) | 13268 | 2725 | 2306 | 1239
months
  Chemotherapy (exclusive): number analyzed (Participants) | 1631 | 1804 | 84 | 75
  Chemotherapy (exclusive) | 5.0 [4.8 to 5.2] | 5.4 [5.1 to 5.8] | 4.4 [3.5 to 5.4] | 4.4 [3.5 to 6.0]
  Endocrine therapy (exclusive): number analyzed (Participants) | 5545 | 0 | 342 | 0
  Endocrine therapy (exclusive) | 12.5 [12.0 to 13.0] |  | 5.9 [5.2 to 7.1] |
  Combination of endocrine therapy and chemotherapy: number analyzed (Participants) | 3383 | 0 | 85 | 0
  Combination of endocrine therapy and chemotherapy | 16.2 [15.4 to 16.7] |  | 9.3 [7.5 to 11.5] |
  Chemotherapy and targeted treatment: number analyzed (Participants) | 699 | 921 | 674 | 1164
  Chemotherapy and targeted treatment | 7.2 [6.7 to 7.8] | 6.5 [6.1 to 6.8] | 9.9 [8.4 to 10.9] | 12.3 [11.3 to 13.0]
  Combination of endocrine therapy and targeted treatment: number analyzed (Participants) | 492 | 0 | 85 | 0
  Combination of endocrine therapy and targeted treatment | 19.4 [15.7 to 23.1] |  | 12.2 [9.9 to 15.8] |
  Combination of chemotherapy, endocrine therapy and targeted treatment: number analyzed (Participants) | 1518 | 0 | 1036 | 0
  Combination of chemotherapy, endocrine therapy and targeted treatment | 14.5 [13.8 to 15.1] |  | 24.6 [22.8 to 27.0] |

3. Secondary Outcome: Association Between Overall Survival and Real-world Progression-free Survival for Commonly Prescribed First-line Treatment Strategies
Description: Individual-level association between rwPFS and OS estimated using a Spearman rank correlation coefficient.
Time Frame: 10 years
Population: Individual-level association between rwPFS and OS is reported for major combinations of treatments.
  For the combination "OTHER", this individual-level association is not reported given the populations are highly heterogeneous, and therefore reporting ondividual-level association is not clinically relevant.
  When the number of participants in a row is "0", this means that the combinbation of treatments (defined by the row) was provided to 0 woman of the population (defined by the column).
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Women With a Diagnosis of HR+ /HER2- Metastatic Breast Cancer (mBC) | Women With a Diagnosis of HR- /HER2- Metastatic Breast Cancer (mBC) | Women With a Diagnosis of HR+ /HER2+ Metastatic Breast Cancer (mBC) | Women With a Diagnosis of HR- /HER2+ Metastatic Breast Cancer (mBC)
Number analyzed (Participants) | 13268 | 2725 | 2306 | 1239
Correlation coefficient
  Chemotherapy (exclusive): number analyzed (Participants) | 1631 | 1804 | 84 | 75
  Chemotherapy (exclusive) | 0.58 [0.54 to 0.61] | 0.81 [0.79 to 0.82] | 0.33 [0.12 to 0.52] | 0.67 [0.51 to 0.78]
  Endocrine therapy (exclusive): number analyzed (Participants) | 5545 | 0 | 342 | 0
  Endocrine therapy (exclusive) | 0.66 [0.64 to 0.68] |  | 0.43 [0.32 to 0.53] |
  Combination of endocrine therapy and chemotherapy: number analyzed (Participants) | 3383 | 0 | 85 | 0
  Combination of endocrine therapy and chemotherapy | 0.78 [0.76 to 0.79] |  | 0.72 [0.58 to 0.82] |
  Chemotherapy and targeted treatment: number analyzed (Participants) | 699 | 921 | 674 | 1164
  Chemotherapy and targeted treatment | 0.45 [0.39 to 0.51] | 0.73 [0.69 to 0.76] | 0.67 [0.61 to 0.72] | 0.81 [0.78 to 0.84]
  Combination of endocrine therapy and targeted treatment: number analyzed (Participants) | 492 | 0 | 228 | 0
  Combination of endocrine therapy and targeted treatment | 0.61 [0.51 to 0.70] |  | 0.71 [0.61 to 0.78] |
  Combination of chemotherapy, endocrine therapy and targeted treatment: number analyzed (Participants) | 1518 | 0 | 1036 | 0
  Combination of chemotherapy, endocrine therapy and targeted treatment | 0.7 [0.67 to 0.73] |  | 0.78 [0.74 to 0.82] |

ADVERSE EVENTS:
Time Frame: Adverse events were not collected for this study.
Description: Adverse events were not collected for this study.
Arm/Group | Women With a Diagnosis of HR+ /HER2- Metastatic Breast Cancer (mBC) | Women With a Diagnosis of HR- /HER2- Metastatic Breast Cancer (mBC) | Women With a Diagnosis of HR+ /HER2+ Metastatic Breast Cancer (mBC) | Women With a Diagnosis of HR- /HER2+ Metastatic Breast Cancer (mBC)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT03676257/Prot_SAP_000.pdf